CLINICAL TRIAL: NCT06679660
Title: Anesthetic Effectiveness of Mental/incisive Nerve Block Versus Inferior Alveolar Nerve Block in Mandibular I. and II. Premolars with Symptomatic Irreversible Pulpitis: a Randomized Clinical Trial
Brief Title: Comparative Assessment of Mental/Incisive and Inferior Alveolar Nerve Block Anesthesia in Root Canal Treatment of Mandibular Premolars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Tolga Sulek, Specialist of Endodontics, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023/130/86
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Mandibular Nerve; Mandibular Nerve Blocks; Premolars; Mental Nerve Block
Keywords: Inferior alveolar nerve block; local anesthesia; mental nerve block; pain; premolar
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Pain | interventions — Carticaine

STUDY DESIGN:
Intervention Model Description: Single blinded randomized clinical study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inferior Alveoler Nerve Block (Experimental)
  Interventions: Other: inferior alveolar nerve block with 4% articaine
- Mental/Incisive Nerve Block (Experimental)
  Interventions: Other: Mental/Incisive Nerve Block (%4 Articaine)

INTERVENTIONS:
Other: inferior alveolar nerve block with 4% articaine — A single ampoule of 4% articaine was administered to a cohort of patients presenting with irreversible pulpitis in the first or second mandibular premolars, designated for Inferior Alveolar Block anesthesia via the mandibular foramen.
  Arms: Inferior Alveoler Nerve Block
Other: Mental/Incisive Nerve Block (%4 Articaine) — A single ampoule of 4% articaine was administered to a cohort of patients presenting with irreversible pulpitis in the first or second mandibular premolars, designated for Mental or Incisive Nerve Block anesthesia via the mental foramen.
  Arms: Mental/Incisive Nerve Block

SUMMARY:
The goal of this clinical trial is to systematically compare the pain scores and anesthesia efficacy of IANB and MNB in the treatment of symptomatic mandibular first and second premolars. This study aims to address gaps in current evidence and clarify whether these anesthesia techniques differ in effectiveness and patient experience during endodontic procedures. The hypotheses include: (i) no difference in pain perception between IANB and MNB, (ii) no difference between first and second premolars with IANB, and (iii) no difference between first and second premolars with MNB.

ELIGIBILITY:
Inclusion Criteria:

* Individuals classified as ASA 1 or ASA 2.
* Age range of 18 to 65 years.
* No known allergies to articaine or epinephrine.
* Absence of facial paresthesia.
* No use of analgesic medications within 6 hours prior to treatment.
* No use of medications, such as tricyclic antidepressants or beta blockers, that may interfere with anesthesia.
* No pathological conditions at the planned injection site.
* Periodontal pocket depth of 3 mm or less.
* Mandibular first or second premolars diagnosed with symptomatic irreversible pulpitis.
* Teeth meeting Glickman's gingival health criteria upon periodontal examination.
* Radiographically closed root apex with no detectable pathology.
* Patients must be literate and able to comprehend the use of a pain scale to provide informed consent voluntarily.

Exclusion Criteria:

* Presence of systemic conditions contraindicating endodontic treatment. Age below 18 or above 65 years.
* Pregnancy.
* Documented allergy to articaine with 1:100,000 epinephrine.
* Evidence of periapical pathology or radiolucency observed in radiographs.
* Recent use of central nervous system depressants or analgesic medication within 6 hours prior to treatment.
* Absence of reported lip numbness 10 minutes following IANB or MINB injection. Presence of a large restoration on the affected tooth.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | Following anesthesia administration, a 10-minute waiting period was observed. Patients completed a Numerical Rating Scale immediately upon initiation of the endodontic cavity procedure and again after the start of pulp extirpation.
  The patients were asked to rate the pain experienced during endodontic access cavity preparation and pulp extirpation using a Numerical Rating Scale. The Numerical Rating Scale was printed on A4 paper, scaled to fit horizontally, with values from 0 to 10 displayed along a bar. The Numerical Rating Scale uses a 0 to 10 scale, with increments of one unit. Patients were instructed to mark '0' if they experienced no pain, select a value between "1" and "3" for mild pain, a value between "4" and "6" for moderate pain, and a value between "7" and "10" for severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University Dentistry Faculty Department of Endodontics Clinic, Adana, Turkey (Türkiye)